CLINICAL TRIAL: NCT00333931
Title: Pilot Trial of Neural Correlates of Response to Treatment of PTSD-Associated Impulsive Aggression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: Dr. Thomas A. Kent (Unknown); Dr. Stacey Holmes (Unknown); Dr. Su Bailey (Unknown); Dr. Mark Kunik (Unknown); Dr. Melinda Stanley (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 18342
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2006-06-06 (Estimated); Status verified 2006-06

CONDITIONS: Impulsive Aggression; Posttraumatic Stress Disorder
Keywords: Impulsive Aggression; Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Phenytoin; Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Phenytoin
Behavioral: Cognitive Behavioral Therapy

SUMMARY:
The purpose of this study is to identify changes in brain functioning which are related to reduced frequency and/or intensity of impulsive aggressive actions after treatment of PTSD-related impulsive aggression with either phenytoin or cognitive behavioral therapy.

DETAILED DESCRIPTION:
Objective One: One study objective is to evaluate potential effect sizes of phenytoin and cognitive behavioral therapy for PTSD-related impulsive aggression.

Hypothesis: Phenytoin and cognitive behavioral therapy are hypothesized to be effective in the treatment of PTSD-related impulsive aggression based on studies previously outlined.

Plan: Patients enrolled in this pilot study will be randomized to receive an eight-week course of treatment with phenytoin or cognitive behavioral therapy in the Trauma Recovery Program at the Veterans's Affairs Medical Center in Houston, Texas.

Objective Two: Another study objective is to begin to attempt to delineate potential neural correlates of treatment-related reductions in PTSD-related impulsive aggression.

Hypothesis: Potential neural correlates of treatment-related reduction in intensity and/or severity of impulsive-aggressive acts are hypothesized to include changes in: 1) thalamic activation reflecting more effective thalamic sensory gating, with anticipation of increased activation of the thalamus post-treatment 2) activation of brain regions associated with verbal information processing, with the anticipation of increased activation of these regions post-treatment 3) activation of prefrontal regions, including the anticipation of increased activation of the medial and/or orbital prefrontal cortex post-treatment, 4) amygdalar activation, with the anticipation of decreased activation of the amygdala post-treatment 5) hippocampal activation, with the anticipation of increased activation of the hippocampus post-treatment, and/or, 6) right-left hemispheric dissociation of brain processing of stimuli, with the anticipation of greater degrees of bilaterality of brain processing of stimuli post-treatment. Specifically, greater degrees of activation of left hemispheric brain structures are anticipated in post-treatment fMRI scans.

Plan: Patients with PTSD-associated impulsive aggression will undergo an eight-week course of treatment with phenytoin or CBT. Treatment-related changes in impulsive-aggressive acts will be correlated with changes in brain activation comparing pre- and post-treatment fMRI scans utilizing a standardized Go-No Go task which has been used in the study of impulsive aggressive individuals.

ELIGIBILITY:
Inclusion Criteria:

- Inclusion Criteria for both groups will be right-handed adult combat veterans over the age of 18 who meet criteria for PTSD via Structured Clinical Interview (SCID-I, First, 2002) and Impulsive Aggression as the primary diagnoses. To be included in the study with a designation of Impulsive Aggression, patients must have committed at least three aggressive acts over the preceding three months meeting criteria for impulsive aggressive acts by Impulsive/Premeditated Aggression Scales (IPAS) criteria (Stanford et al 2003) based on a semi-structured interview of the patient and his/her significant other. An impulsive aggressive act is defined as a hair-trigger, non-premeditated response to a stimulus that results in an immediate aggressive act or an agitated state that culminates in an aggressive act, which is clearly disproportionate to the triggering stimulus. Inclusion criteria for both groups also includes the availability for participation of a significant other who can participate in the study. The significant other will need to accompany the study participant to the initial assessment interview and complete measures of aggressive acts which have been committed by the study participants in the three months prior to the start of the study, and aggressive acts during the previous two weeks at two-week interval follow-up visits throughout the eight-week treatment period.

Exclusion Criteria:

* Exclusion Criteria for both groups will include exclusion criteria for MRI scanning, and known claustrophobia requiring sedation in the past during MRI scanning. MRI exclusion criteria will include metallic implants, implanted devices of any kind, such as a cardiac pacemaker, cardiac defibrillator, insulin pump, vagal nerve stimulator, cochlear implant, metallic splinters in the eye, ferromagnetic clips or metal in the head or brain (as from previous injury or head/brain surgery including brain aneurysm clipping), lead wires of any kind, clips or stints anywhere in the body, such as clips for arterial aneurysm clipping, stints in cardiac arteries or other arteries anywhere in the body, prosthetic heart valves, stapedial implants of any kind (implants in the inner ear).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2006-06

PRIMARY OUTCOMES:
change in impulsive aggressive acts measured by OAS-M

SECONDARY OUTCOMES:
change in regional brain activation as measured by FMRI
change in PTSD symptoms as measured by CAPS
change in depression symptoms as measured by BDI

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Kent, MD, Study Director — Veterans Affairs Medical Center-Houston
Locations (1):
- Veterans Affairs Medical Center, Houston, Texas, United States